CLINICAL TRIAL: NCT06606782
Title: Evaluation of Incidence of Stomach Fullness in Elective Surgical Patients and Investigation of Associated Factors: Prospective Observational Study
Brief Title: Incidence of Stomach Fullness and Associated Factors in Elective Surgical Patients
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Başar Erdivanlı, Assoc. Prof., Recep Tayyip Erdogan University
Other Study IDs: 2020/202
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Gastric Emptying; Preoperative Care; Preoperative Fasting; Elective Surgical Procedures; Ultrasonography
Keywords: Gastrointestinal Contents / diagnostic imaging*; Ultrasonography / methods*; Respiratory Aspiration / prevention & control*; Preoperative Care / methods; Risk Factors / evaluation; Patient-Reported Outcomes / methods; Humans
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Elective Surgery Patients: This cohort includes adult patients undergoing elective surgery who were assessed for residual gastric content using ultrasound and a preoperative questionnaire. All patients adhered to standard preoperative fasting guidelines prior to the assessment.

SUMMARY:
The aim of this prospective, observational study is to evaluate the incidence of residual gastric content in elective surgical patients who adhered to preoperative fasting guidelines and to investigate associated patient-related factors. Ultrasound (USG) has been identified as a valuable tool for assessing residual gastric content, and this study compares its efficacy against traditional questionnaire-based predictions. The study also examines the practicality and accuracy of different gastric volume estimation formulas and evaluates their correlation with aspiration risk.

A total of 475 patients were enrolled in the study, of whom 404 completed both the questionnaire and USG examination. All participants were adult patients scheduled for elective surgery, following standard fasting protocols. The ultrasound examination assessed the presence of solid or fluid content in the stomach, and patients were classified according to qualitative Perlas risk scores (Grade 0: Low, Grade 1: Moderate, Grade 2: High risk of aspiration). The questionnaire collected patient-reported factors, such as symptoms of early satiety, history of cholelithiasis, and comorbidities like diabetes or chronic obstructive pulmonary disease (COPD).

The primary objective of this study was to evaluate the efficacy of USG in detecting residual gastric content and compare it with questionnaire-based risk predictions. Logistic regression analysis identified early satiety and cholelithiasis as significant predictors of a full stomach and higher aspiration risk. Fasting duration was found to have a protective effect, reducing the likelihood of a full stomach. While many patient characteristics traditionally associated with delayed gastric emptying, such as age and diabetes, did not significantly correlate with the outcomes, early satiety and cholelithiasis proved to be key factors influencing gastric content.

In addition, this study explored the performance of several gastric volume estimation formulas, including the Michiko, Bouvet, and Perlas 2019/2020 formulas. The findings indicated significant limitations in these formulas, with many patients being estimated to have negative gastric volumes, particularly by the Michiko and two of Perlas' formulas. This highlights the inadequacies of current formulas in accurately predicting gastric volume, necessitating further refinement and development of new models that better account for physiological variability.

Furthermore, the agreement between questionnaire-based predictions and USG findings was assessed using Cohen's Kappa, which indicated fair agreement (Kappa value = 0.282). This suggests that while the questionnaire can serve as a screening tool to identify patients at risk of aspiration, it cannot replace the accuracy and reliability of USG in clinical practice.

Secondary objectives of the study included comparing the time-efficiency and ease of implementation between USG and the questionnaire-based assessments. USG proved to be more time-efficient, taking an average of 2.5 minutes per examination, compared to 3-5 minutes for completing the questionnaire. This speed, combined with its objective nature, underscores USG's value as a practical tool in the preoperative setting.

In conclusion, USG was found to be an effective and efficient tool for assessing residual gastric content and predicting aspiration risk, outperforming traditional questionnaire-based assessments. The inadequacy of current gastric volume estimation formulas points to the need for further research to develop more accurate and context-specific assessment tools. Comprehensive preoperative evaluation incorporating USG and patient-reported symptoms may improve patient safety by reducing the risk of aspiration during elective surgery.

DETAILED DESCRIPTION:
This study is a prospective observational research project designed to evaluate the incidence of residual gastric content in patients scheduled for elective surgery and to investigate patient-related factors that influence gastric emptying. The study primarily employs ultrasonography (USG) as a tool for assessing the presence of residual gastric content and compares its efficacy with traditional questionnaire-based assessments. Additionally, the study examines the utility and accuracy of various gastric volume estimation formulas, assessing their correlation with observed gastric content and aspiration risk.

Study Design:

Participants were enrolled based on pre-defined inclusion and exclusion criteria, including adult patients scheduled for elective surgery who adhered to standard preoperative fasting guidelines. Following a detailed informed consent process, patients were asked to complete a preoperative questionnaire, which gathered data on demographic characteristics, medical history, and patient-reported symptoms, such as early satiety, history of cholelithiasis, and other relevant comorbidities. Ultrasound examinations were performed by a single trained investigator to ensure consistency in imaging and interpretation.

USG was utilized to assess residual gastric content, including both solid and fluid content. The antrum cross-sectional area was measured in the supine and right lateral decubitus positions, and gastric volume was estimated using four different formulas: Michiko, Bouvet, two fo Perlas' formulas developed in differnet investigations. Patients were classified into three groups according to the Perlas risk score, which is based on ultrasound findings of gastric content (Grade 0 = low risk, Grade 1 = moderate risk, Grade 2 = high risk of aspiration). The primary outcome was the identification of a full stomach, defined as the presence of solid content or fluid contentbased on ultrasound findings.

Registry Procedures and Quality Control:

Quality assurance procedures were integrated into the study to ensure the reliability of both questionnaire-based data and ultrasound findings. The following processes were implemented:

1. Data Validation: All questionnaire responses and ultrasound measurements were reviewed for consistency and completeness. In the event of data entry errors or inconsistencies, the original data sources (questionnaires or ultrasound logs) were consulted for clarification and correction.
2. Source Data Verification: Ultrasound findings were periodically cross-referenced with patient charts and medical records to verify the accuracy of reported comorbidities and other patient characteristics.
3. Data Dictionary and Coding: The study utilized a detailed data dictionary for all variables, including categorical coding for risk factors, comorbidities, and ultrasound findings. For example, the World Health Organization's MedDRA coding was used for medical conditions, and normal ranges for fasting times and antrum cross-sectional area were predefined based on existing literature.
4. Standard Operating Procedures (SOPs): SOPs were developed for patient recruitment, ultrasound measurements, data collection, data management, and data analysis. These procedures included regular checks for missing or incomplete data, predefined criteria for image quality in ultrasound readings, and protocols for identifying and addressing any out-of-range results.

Sample Size Assessment:

A sample size of 207 patients was calculated using the G-Power program (version 3.1.9.7), with the degrees of freedom set to 3 and an effect size of 0.3. This sample size was based on examining two patient groups with a categorical variable containing four categories, with a type I error rate of 0.05 and a type II error rate of 0.1. To account for subgroup analyses and potential registration errors, a target of at least 300 patients was set. The final number of patients completing both the questionnaire and ultrasound was 404.

Plan for Missing Data:

To address missing data, the following strategies were implemented:

* Any incomplete questionnaire responses were flagged, and patients were contacted to complete the missing information, where possible.
* Missing ultrasound measurements were rare, but if ultrasound images were deemed inadequate (e.g., poor image quality or patient inability to tolerate positioning), these patients were excluded from the specific analyses.
* For missing or inconsistent values, a complete-case analysis was employed, excluding individuals from specific models if key variables were not available.
* Sensitivity analyses were conducted to assess the impact of missing data on the final results.

Statistical Analysis Plan:

Data analysis was conducted using R statistical software (version 4.1.2). Statistical techniques were selected based on the study objectives:

1. Primary Objective (USG Efficacy):

   * Logistic regression models were employed to assess the relationship between patient characteristics (e.g., early satiety, cholelithiasis) and full stomach based on USG findings. The dependent variable was the binary outcome of full stomach vs. empty stomach.
   * Qualitative scoring based on the Perlas risk score was incorporated to evaluate aspiration risk, with separate logistic models developed to predict Grade 0 (low risk), Grade 1 (moderate risk), and Grade 2 (high risk).
   * Model performance was assessed using the area under the receiver operating characteristic (ROC) curve (AUC), and the optimal cutoff points were determined using Youden's index to balance sensitivity and specificity.
2. Secondary Objective (Questionnaire vs. USG):

   * Cohen's Kappa statistic was used to assess agreement between questionnaire-based predictions and USG findings. This analysis aimed to determine how well the questionnaire could predict residual gastric content and aspiration risk compared to USG.
   * Time-efficiency was analyzed by comparing the average duration of completing the questionnaire (3-5 minutes) vs. the ultrasound examination (2.5 minutes).
3. Gastric Volume Estimation Formulas:

   * Correlation coefficients (Spearman's rank) were calculated to determine the association between estimated gastric volumes from the four formulas (Michiko, Bouvet, two of Perlas' formulas) and the ultrasound findings (full stomach and aspiration risk).
   * Logistic regression models were developed to evaluate whether the estimated gastric volumes from each formula were significant predictors of full stomach or aspiration risk. Negative or non-significant results were flagged as indicators of formula limitations.
4. Adjusted Models:

   * Multivariate models adjusting for potential confounders (e.g., age, sex, comorbidities such as diabetes) were developed to ensure that observed associations between patient characteristics and gastric content or risk were not confounded by other variables.
   * A complete-case analysis was performed for all multivariate models, excluding patients with missing values for any of the key variables.

Limitations:

The study acknowledges several limitations. First, no direct measurement of gastric volume was obtained through orogastric tube aspiration, limiting the ability to definitively compare USG findings to a gold standard. Second, the analysis was constrained by the relatively small number of patients (n = 57) for whom volume estimation was possible, particularly due to negative or invalid results from the gastric volume formulas. Lastly, the study was performed in a single center, and all ultrasound measurements were conducted by a single investigator, which, while minimizing inter-operator variability, may limit the generalizability of the findings to other settings.

Future Directions:

Future studies should focus on refining the gastric volume estimation formulas and exploring additional patient-reported symptoms and clinical factors that may affect gastric emptying. There is also a need to standardize ultrasound protocols and validate the findings in a multi-center, diverse patient population. In addition, comparisons with other preoperative risk assessment tools, such as orogastric tube suction, should be explored.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective surgery
* adhered to preoperative fasting guidelines
* provided written informed consent

Exclusion Criteria:

* children under 18 years of age
* pregnant women
* patients requiring emergency surgery
* patients with a history of previous stomach surgery
* patients who did not complete the sufficient fasting period (less than 8 hours)
* patients with whom reliable cooperation for questionnaire completion could not be established (e.g., inability to provide reliable answers)
* patients who could not be positioned on their right side due to clinical conditions
* patients in whom sufficient quality imaging of the gastric antrum could not be obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery at the Recep Tayyip Erdoğan University Faculty of Medicine Rize Training and Research Hospital
Sampling Method: Non-Probability Sample
Enrollment: 404 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Full Stomach in Elective Surgical Patients as Assessed by Ultrasound | At the time of preoperative assessment, within 2 hours prior to surgery.
  The number of participants with full stomachs, as determined by the presence of solid content or fluid content using preoperative gastric ultrasound. Full stomach is defined as either solid content or clear fluid in the supine or right lateral decubitus positions.

SECONDARY OUTCOMES:
Correlation Between Preoperative Fasting Duration and Incidence of Full Stomach as Assessed by Ultrasound | At the time of preoperative assessment, within 2 hours prior to surgery.
  The correlation between the duration of preoperative fasting and the likelihood of having a full stomach, as determined by gastric ultrasound. Fasting duration is self-reported by participants and compared with ultrasound findings.
Perlas Risk Score for Aspiration Risk as Assessed by Ultrasound | At the time of preoperative assessment, within 2 hours prior to surgery.
  The number of participants stratified into low, moderate, or high aspiration risk groups based on the Perlas qualitative risk scoring system. The Perlas score is based on the gastric content identified via ultrasound, with Grade 0 indicating empty stomach, Grade 1 indicating clear fluid only in right lateral decubitus position but no solid content or fluid &amp;amp;amp;gt; 1.5 mL/kg, and Grade 2 indicating solid content or clear fluid in both the supine and right lateral decubitus positions, or fluid volume &amp;amp;gt; 1.5 mL/kg
Agreement Between Questionnaire-Based Risk Prediction and Ultrasound Findings for Aspiration Risk | At the time of preoperative assessment, within 2 hours prior to surgery.
  ultrasound findings, as measured by Cohen's Kappa statistic. The questionnaire assesses patient-reported risk factors such as early satiety, while ultrasound is used to detect full stomachs and quantify the aspiration risk.
Time Efficiency of Ultrasound vs. Questionnaire-Based Gastric Content Assessment | At the time of preoperative assessment, within 2 hours prior to surgery.
  The time required to complete ultrasound-based gastric content assessment compared to questionnaire-based risk factor collection. The time taken for each method will be recorded and compared for efficiency.
Gastric Volume Estimation Using Multiple Formulae and Correlation with Aspiration Risk | At the time of preoperative assessment, within 2 hours prior to surgery.
  Estimated gastric volumes derived from four different formulas (Michiko, Bouvet, two formulas from Perlas) based on ultrasound measurements. The relationship between estimated gastric volume and aspiration risk (as assessed by Perlas risk score) will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdoğan University Rize Training and Research Hospital, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Only the Individual Patient Data (IPD) included in the final results publication will be shared. Records from patients who were excluded due to incomplete data-such as those unable to complete either the questionnaire or the ultrasound examination, as specified in the exclusion criteria-have been omitted from the digital dataset used for analysis. These records were not used in the final results to ensure the accuracy and integrity of the findings.
Supporting Information: CSR, Analytic Code
Time Frame: Starting at January 2025, the IPD and analytical code will be shared.
Access Criteria: Individual patient data (IPD) and/or analytical code may be shared upon request from researchers affiliated with recognized academic or research institutions, provided they have a valid organizational email address. Requests must include the name of the Ethics Committee, decision number, and date of approval.
  Sharing of data will be limited to de-identified and anonymized datasets to protect patient confidentiality. To further ensure patient privacy, informed consents will not be shared directly with individual researchers but may be reviewed by accredited institutions or journals for verification purposes. Data sharing will only be allowed for purposes such as systematic reviews, meta-analyses, or reanalysis of study findings, where the intent is to advance scientific knowledge while preserving the confidentiality of patient participants.

REFERENCES:
- [Background] Sugita M, Matsumoto M, Tsukano Y, Fukunaga C, Yamamoto T. Gastric emptying time after breakfast in healthy adult volunteers using ultrasonography. J Anesth. 2019 Dec;33(6):697-700. doi: 10.1007/s00540-019-02694-6. Epub 2019 Oct 19. PMID 31630260
- [Background] Bouvet L, Mazoit JX, Chassard D, Allaouchiche B, Boselli E, Benhamou D. Clinical assessment of the ultrasonographic measurement of antral area for estimating preoperative gastric content and volume. Anesthesiology. 2011 May;114(5):1086-92. doi: 10.1097/ALN.0b013e31820dee48. PMID 21364462
- [Background] Perlas A, Davis L, Khan M, Mitsakakis N, Chan VW. Gastric sonography in the fasted surgical patient: a prospective descriptive study. Anesth Analg. 2011 Jul;113(1):93-7. doi: 10.1213/ANE.0b013e31821b98c0. Epub 2011 May 19. PMID 21596885
- [Background] Perlas A, Mitsakakis N, Liu L, Cino M, Haldipur N, Davis L, Cubillos J, Chan V. Validation of a mathematical model for ultrasound assessment of gastric volume by gastroscopic examination. Anesth Analg. 2013 Feb;116(2):357-63. doi: 10.1213/ANE.0b013e318274fc19. Epub 2013 Jan 9. PMID 23302981
- [Background] Bouvet L, Desgranges FP, Aubergy C, Boselli E, Dupont G, Allaouchiche B, Chassard D. Prevalence and factors predictive of full stomach in elective and emergency surgical patients: a prospective cohort study. Br J Anaesth. 2017 Mar 1;118(3):372-379. doi: 10.1093/bja/aew462. PMID 28203726
- [Background] Perlas A, Arzola C, Van de Putte P. Point-of-care gastric ultrasound and aspiration risk assessment: a narrative review. Can J Anaesth. 2018 Apr;65(4):437-448. doi: 10.1007/s12630-017-1031-9. Epub 2017 Dec 11. PMID 29230709
- [Background] El-Boghdadly K, Wojcikiewicz T, Perlas A. Perioperative point-of-care gastric ultrasound. BJA Educ. 2019 Jul;19(7):219-226. doi: 10.1016/j.bjae.2019.03.003. Epub 2019 Apr 24. No abstract available. PMID 33456894
- [Background] Goyal RK, Cristofaro V, Sullivan MP. Rapid gastric emptying in diabetes mellitus: Pathophysiology and clinical importance. J Diabetes Complications. 2019 Nov;33(11):107414. doi: 10.1016/j.jdiacomp.2019.107414. Epub 2019 Aug 8. PMID 31439470
- [Background] Zhou L, Yang Y, Yang L, Cao W, Jing H, Xu Y, Jiang X, Xu D, Xiao Q, Jiang C, Bo L. Point-of-care ultrasound defines gastric content in elective surgical patients with type 2 diabetes mellitus: a prospective cohort study. BMC Anesthesiol. 2019 Oct 10;19(1):179. doi: 10.1186/s12871-019-0848-x. PMID 31601180
- [Background] Chang JE, Kim H, Won D, Lee JM, Jung JY, Min SW, Hwang JY. Ultrasound assessment of gastric content in fasted patients before elective laparoscopic cholecystectomy: a prospective observational single-cohort study. Can J Anaesth. 2020 Jul;67(7):810-816. doi: 10.1007/s12630-020-01668-7. Epub 2020 Apr 20. PMID 32314262
- [Background] Nguyen L, Wilson LA, Miriel L, Pasricha PJ, Kuo B, Hasler WL, McCallum RW, Sarosiek I, Koch KL, Snape WJ, Farrugia G, Grover M, Clarke J, Parkman HP, Tonascia J, Hamilton F, Abell TL; NIDDK Gastroparesis Clinical Research Consortium (GpCRC). Autonomic function in gastroparesis and chronic unexplained nausea and vomiting: Relationship with etiology, gastric emptying, and symptom severity. Neurogastroenterol Motil. 2020 Aug;32(8):e13810. doi: 10.1111/nmo.13810. Epub 2020 Feb 15. PMID 32061038
- [Background] Syed AR, Wolfe MM, Calles-Escandon J. Epidemiology and Diagnosis of Gastroparesis in the United States: A Population-based Study. J Clin Gastroenterol. 2020 Jan;54(1):50-54. doi: 10.1097/MCG.0000000000001231. PMID 31135630
- [Background] Goyal RK. Gastric Emptying Abnormalities in Diabetes Mellitus. N Engl J Med. 2021 May 6;384(18):1742-1751. doi: 10.1056/NEJMra2020927. No abstract available. PMID 33951363
- [Background] Shaw M, Waiting J, Barraclough L, Ting K, Jeans J, Black B; Pan-London Peri-operative Audit and Research Network. Airway events in obese vs. non-obese elective surgical patients: a cross-sectional observational study. Anaesthesia. 2021 Dec;76(12):1585-1592. doi: 10.1111/anae.15513. Epub 2021 Jun 22. PMID 34156711
- [Background] Sun J, Wei G, Hu L, Liu C, Ding Z. Perioperative pulmonary aspiration and regurgitation without aspiration in adults: a retrospective observational study of 166,491 anesthesia records. Ann Palliat Med. 2021 Apr;10(4):4037-4046. doi: 10.21037/apm-20-2382. Epub 2021 Mar 23. PMID 33832306
- [Background] Warner MA, Meyerhoff KL, Warner ME, Posner KL, Stephens L, Domino KB. Pulmonary Aspiration of Gastric Contents: A Closed Claims Analysis. Anesthesiology. 2021 Aug 1;135(2):284-291. doi: 10.1097/ALN.0000000000003831. PMID 34019629
- [Background] Assmus F, Hoglund RM, Monnot F, Specht S, Scandale I, Tarning J. Drug development for the treatment of onchocerciasis: Population pharmacokinetic and adverse events modeling of emodepside. PLoS Negl Trop Dis. 2022 Mar 10;16(3):e0010219. doi: 10.1371/journal.pntd.0010219. eCollection 2022 Mar. PMID 35271567
- [Background] Frykholm P, Disma N, Andersson H, Beck C, Bouvet L, Cercueil E, Elliott E, Hofmann J, Isserman R, Klaucane A, Kuhn F, de Queiroz Siqueira M, Rosen D, Rudolph D, Schmidt AR, Schmitz A, Stocki D, Sumpelmann R, Stricker PA, Thomas M, Veyckemans F, Afshari A. Pre-operative fasting in children: A guideline from the European Society of Anaesthesiology and Intensive Care. Eur J Anaesthesiol. 2022 Jan 1;39(1):4-25. doi: 10.1097/EJA.0000000000001599. PMID 34857683